CLINICAL TRIAL: NCT03714035
Title: Measurement of Mandibular Radio Morphometric Indices in Egyptian Population at Different Ages Using Cone Beam Computed Tomography: A Cross Sectional Study
Brief Title: Measurement of Mandibular Radio Morphometric Indices in Egyptian Population at Different Ages
Acronym: Indices
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanaa Sayed Mansy, demonstrator at faculty of dentistry cairo university, Cairo University
Other Study IDs: Hphd; FDCU (Other: faculty of dentistry)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
this study aims to correlate mandibular indices and different ages in a sample of Egyptian population.

DETAILED DESCRIPTION:
this study is an observational cross sectional study to correlate the mandibular radiomorphometric indices with age in sample of egyptian population using CBCT scans at faculty of dentistry cairo university

ELIGIBILITY:
Inclusion Criteria:

* Egyptian individuals with different ages starting from 10 - 70 years.
* Females and males of the mentioned ages.

Exclusion Criteria:

* Individuals younger than 10 and older than 70 years old.
* Presence of a large pathological lesions in the mandible at the areas intended for measurements.
* Patients of severely resorbed mandibular bone.
* Patients with any bony deformity at the inferior border of the mandible.
* Patients with fracture at the areas to be examined.
* Patients with evident radiographic asymmetry.
* Patients with evident radiographic abnormality suggestive of systemic disease predisposing to osteoporosis.
* Patients with current postoperative surgical defect healing at the areas intended for measurements.
* Patients with mandibular reconstruction

Ages: 10 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: a sample of egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
panoramic mandibular index | 2018-2020
  ratio between the thickness of the mandible at the mental foramen area and the distance measured from the inferior border of the mental foramen to the inferior border of the mandible. The value of 0.3 will be considered as normal value while the lower value indicate abnormal inferior border thickness

CONTACTS AND LOCATIONS:
Overall Officials: Dentistry Cairo, Univeristy, Study Chair — Ethical committee faculty if dentustry cairo unveristry
Locations (1):
- Faculty of dentistry cairo univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No